CLINICAL TRIAL: NCT01813981
Title: The Effect of High and Low Roasted Coffee on Vascular Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: COFF2011
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High roast coffee (Placebo Comparator): 110mg caffeine with 108 mg chlorogenic acid at start of study
  Interventions: Dietary Supplement: Control (Caffeine dissolved in water)
- Low roast coffee (Active Comparator): 110 mg caffeine with 235 mg chlorogenic acid at start of the study
  Interventions: Dietary Supplement: Low roast coffee
- Control (Placebo Comparator): 110 mg caffeine at start of study
  Interventions: Dietary Supplement: High roast coffee

INTERVENTIONS:
Dietary Supplement: Low roast coffee — Instant coffee
  Arms: Low roast coffee
Dietary Supplement: High roast coffee — Instant coffee
  Arms: Control
Dietary Supplement: Control (Caffeine dissolved in water) — Caffeine dissolved in water
  Arms: High roast coffee

SUMMARY:
Evidence suggests that a diet rich in plant phenolic compounds may induce beneficial vascular effects. Coffee is a good source of phenolic compounds called chlorogenic acids (CGA), however the level of CGA is reduced during the roasting process.

The aim of this study is to investigate the effect of coffee roasting on vascular response. The investigators hypothesize that coffee roasted to a lesser extent will exert a favourable vascular response over more heavily roasted coffee due to the higher levels of CGA.

ELIGIBILITY:
Inclusion Criteria:

* Male
* A signed consent form
* Age 19-35 years
* Body mass index - 18.5-30 kg/m2
* Normal blood pressure at screening (< 150/90)

Exclusion Criteria:

* Blood pressure > 150/90 mmHg
* Haemoglobin (anaemia marker) < 125 g/l
* Gamma GT (liver enzymes) > 80 IU/l
* Cholesterol > 6.5 mmol/l
* Had suffered a myocardial infarction or stroke in the previous 12 months
* Suffers from any reproductive disorder
* Suffers from any blood-clotting disorder
* Suffers from any metabolic disorders (e.g. diabetes or any other endocrine or liver diseases)
* Any dietary restrictions or on a weight reducing diet
* Drinking more than 21 units per week
* On any lipid-modifying medication
* On any blood pressure lowering medication
* On any medication affecting blood clotting
* Planning on altering consumption of vitamin supplements/fish oil capsules during the course of the study
* Regular or vigorous exercise (3 times/week, 20 minutes each session)
* Smoking
* Vegetarians or vegans

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Vascular response measured by flow mediated dilatation (FMD) | Change from baseline to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, Principal Investigator — University of Reading
Locations (2):
- United Kingdom (2):
  - Department of Food and Nutritional Sciences, Reading, Berkshire
  - University of Reading, Reading, England

REFERENCES:
- [Derived] Mills CE, Flury A, Marmet C, Poquet L, Rimoldi SF, Sartori C, Rexhaj E, Brenner R, Allemann Y, Zimmermann D, Gibson GR, Mottram DS, Oruna-Concha MJ, Actis-Goretta L, Spencer JPE. Mediation of coffee-induced improvements in human vascular function by chlorogenic acids and its metabolites: Two randomized, controlled, crossover intervention trials. Clin Nutr. 2017 Dec;36(6):1520-1529. doi: 10.1016/j.clnu.2016.11.013. Epub 2016 Nov 30. PMID 28012692